CLINICAL TRIAL: NCT07372170
Title: Real-world Observational Study to Evaluate the Effectiveness and Safety of Direct Oral Anticoagulants Compared With Vitamin K Antagonists for Secondary Thrombosis Prevention in Low-risk Thrombotic Antiphospholipid Syndrome Patients
Brief Title: Observational Study to Evaluate the Effectiveness of DOACS for Secondary Thrombosis Prevention in Low-risk Thrombotic APS Patients
Acronym: DOACS-APS
Status: Recruiting | Type: Observational
Sponsor: Infanta Leonor University Hospital (Other)
Collaborators: pInvestiga (Unknown)
Responsible Party: Principal Investigator, Anabel Franco Moreno, Principal Investigator, Infanta Leonor University Hospital
Other Study IDs: DOACS-APS
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Antiphospholipid Syndrome (APS); Venous Thrombosis (Disorder); Thrombophilia
Keywords: Direct oral anticoagulants; Vitamin K antagonists; Low-risk antiphospholipid syndrome; Secondary thrombosis prevention; Real-world study; Observational study; Venous Thrombosis; Antiphospholipid Antibody Profile
MeSH Terms: conditions — Antiphospholipid Syndrome; Venous Thrombosis; Thrombophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with low-risk thrombotic antiphospholipid syndrome receiving direct oral anticoagulants: Patients with low-risk thrombotic antiphospholipid syndrome receiving direct oral anticoagulants for secondary prevention of venous thrombosis according to routine clinical practice. Treatment choice is made by the treating physician, with no intervention
- Patients with low-risk thrombotic antiphospholipid syndrome receiving vitamin K antagonist: Patients with low-risk thrombotic antiphospholipid syndrome receiving vitamin K antagonists for secondary prevention of venous thrombosis according to routine clinical practice. Treatment choice is made by the treating physician, with no intervention

SUMMARY:
This is an observational study designed to evaluate the effectiveness and safety of direct oral anticoagulants (DOACs) compared with vitamin K antagonists (VKAs) for the secondary prevention of thrombosis in patients with low-risk thrombotic antiphospholipid syndrome.

Antiphospholipid syndrome is an autoimmune disorder associated with an increased risk of thrombotic events. Although VKAs have traditionally been the standard treatment, DOACs are increasingly used in clinical practice in selected patients, despite limited evidence in this setting.

This study includes patients with previous venous thrombosis and a low-risk serological profile who are treated with either DOACs or VKAs according to routine clinical practice. The primary objective is to compare thrombotic recurrence and bleeding events between both treatment strategies.

The results of this study will contribute to improving knowledge about the use of DOACs in patients with low-risk thrombotic antiphospholipid syndrome.

DETAILED DESCRIPTION:
Antiphospholipid syndrome (APS) is an autoimmune disorder characterized by the occurrence of arterial, venous, or small-vessel thrombosis in the presence of persistent antiphospholipid antibodies. Patients with thrombotic APS have a high risk of recurrent thrombosis and require long-term anticoagulation. Vitamin K antagonists (VKAs) have traditionally been the treatment of choice in this population.

Direct oral anticoagulants (DOACs) have demonstrated efficacy and safety in other clinical settings, such as venous thromboembolism and non-valvular atrial fibrillation. However, their use in APS remains controversial following randomized clinical trials that showed an increased risk of arterial thrombotic events, particularly in patients with high-risk serological profiles.

Current clinical guidelines suggest that DOACs may be considered in selected patients with low-risk thrombotic APS, defined by venous thrombosis and the absence of triple antiphospholipid antibody positivity. Nevertheless, evidence supporting their use in this specific subgroup is limited.

This observational, analytical, ambispective (retrospective and prospective) study aims to evaluate the effectiveness and safety of DOACs compared with VKAs in patients with low-risk thrombotic APS under routine clinical practice conditions.

Adult patients with a diagnosis of low-risk thrombotic APS who are receiving treatment with DOACs or VKAs at the time of inclusion will be eligible. Anticoagulant therapy will be prescribed at the discretion of the treating physician, with no intervention by the study protocol.

The primary objective is to assess a combined effectiveness and safety endpoint, including thrombotic recurrence and major or clinically relevant bleeding. Secondary objectives include all-cause mortality, cardiovascular mortality, and treatment-related quality of life assessed using the Anti-Clot Treatment Scale (ACTS).

The study will be conducted in Internal Medicine units across Spain and is expected to provide relevant real-world evidence to support clinical decision-making in the anticoagulant management of patients with low-risk thrombotic antiphospholipid syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with a diagnosis of thrombotic antiphospholipid syndrome.
* Low-risk antiphospholipid syndrome defined by previous venous thrombosis and a single or double positive antiphospholipid antibody profile (lupus anticoagulant, anticardiolipin antibodies, and/or anti-beta-2-glycoprotein I antibodies).
* Patients receiving long-term anticoagulant treatment with direct oral anticoagulants or vitamin K antagonists according to routine clinical practice.
* At least 2 weeks of continuous anticoagulant treatment before study inclusion.

Exclusion Criteria:

* Age <18 years.
* Triple antiphospholipid antibody positivity.
* History of arterial thrombosis.
* Anticoagulation for indications other than secondary prevention of venous thrombosis related to antiphospholipid syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients with low-risk thrombotic antiphospholipid syndrome managed in routine clinical practice at Internal Medicine units in Spain. Eligible patients have a history of venous thrombotic events and a low-risk antiphospholipid antibody profile and are treated with either direct oral anticoagulants or vitamin K antagonists at the discretion of the treating physician. The study combines retrospective and prospective data collection and does not involve any intervention beyond standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of recurrent venous thrombosis | 24 months
  Occurrence of recurrent venous thrombosis during follow-up.

OTHER OUTCOMES:
Major or clinically relevant non-major bleeding | 24 months
  Occurrence of major bleeding or clinically relevant non-major bleeding events during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Anabel Franco-Moreno, MD, PhD, Principal Investigator — Sociedad Española De Medicina Interna
Locations (2):
- Spain (2):
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
  - Hospital Universitario Infanta Sofía, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in publications arising from this study will be made available upon reasonable request. Data will be shared after publication of the primary results, subject to approval by the study investigators and in accordance with applicable ethical and legal requirements. Requests must include a methodologically sound research proposal, and data will be provided under a data sharing agreement to ensure participant confidentiality.